CLINICAL TRIAL: NCT07306572
Title: Comparative Study Between Loupe-Assisted Varicocelectomy With Nitroglycerin Instillation Versus Microscopic Varicocelectomy
Brief Title: Loupe-Assisted Varicocelectomy With Nitroglycerin Instillation Versus Microscopic Varicocelectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Dogha, assistant professor of urology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-652
Record Dates: First submitted 2025-11-21; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Nitroglycerine Instillation in Loop-assisted Varicocelectomy; Microscopic Varicocelectomy
Keywords: loop-assisted; microscopic; varicocelectomy; nitroglycerine

STUDY DESIGN:
Intervention Model Description: group A where we use nitroglycerine instillation with loop-assisted varicocelectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- loop-assisted varicocelectoy with nitroglycerin instillation group (Experimental): Varicocelectomy is done using loop to improve vision and nitroglycerine instillation to cause vessel dilation and improve identification of arteries to avoid injury
  Interventions: Procedure: loop-assisted varicocelectomy with nitroglycerine instillation
- microscopic varicocelectomy group (Active Comparator): varicocelectomy done using microscopic assistance to improve vision
  Interventions: Procedure: microscopic varicocelectomy

INTERVENTIONS:
Procedure: loop-assisted varicocelectomy with nitroglycerine instillation — nitroglycerine instillation with loop-assisted varicocelectomy
  Arms: loop-assisted varicocelectoy with nitroglycerin instillation group
Procedure: microscopic varicocelectomy — we use microscopic magnification in varicocelectomy
  Arms: microscopic varicocelectomy group

SUMMARY:
Goal: To evaluate the safety and effectiveness of subinguinal microscopic varicocelectomy versus subinguinal loupe-assisted varicocelectomy with nitroglycerin instillation as a vasodilator.

Materials and Procedures: 60 patients were enrolled in our prospective randomized trial between May 2023 and April 2024. They were split into two groups, Group A undergoing Loupe varicocelectomy (LV) with nitroglycerin instillation, and Group B undergoing Microscopic varicocelectomy (MV). Nitroglycerin was administered to the LV group following delivery and cord incision to help visualize cord veins and arterial pulse and avoid confusion with other cord structures that were to be preserved. Three months after the procedure, both groups had scrotal Doppler and semen analysis.

DETAILED DESCRIPTION:
Introduction:

The dilation and anomaly of the testicular veins within the spermatic cord is known as varicocele. It is the most frequent treatable cause of male infertility and a significant contributor to poor spermatogenesis. Only 20% of males with verified varicocele, according to reports, have infertility issues . Disrupting the venous return from the pampiniform plexus's enlarged veins is the main objective of varicocele repair. The internal spermatic artery, vas deferens, and spermatic cord lymphatics are among the vital spermatic cord structures that must be preserved during surgery .

Urologists now use a variety of techniques for varicocele repair, such as inguinal, subinguinal, retroperitoneal, laparoscopic, angioembolization, and both loupe-assisted (LV) and microscopic varicocelectomy (MV) .

The results of varicocelectomy have been greatly improved by the use of surgical microscopes and loupes, and MV is now regarded as the gold standard procedure. Recurrence rates and the frequency of problems such hydrocele formation are remarkably low when done with the right expertise and experience, ranging from 1-2% and 0-1%, respectively.Vasodilators have been used in certain cases to increase vein recognition and visualize the pulse of the testicular artery during surgery, which may further improve surgical outcomes and lower complications .Compared to surgical microscopes, surgical loupes are more widely available, less expensive, and have a simpler learning curve .

Patient and methods:

After receiving clearance from the Fayoum Faculty of Medicine's ethics committee (Number -M 652) in May 2023, this study included 60 patients who were admitted to the urology department of Fayoum University Hospital and had been diagnosed with clinical varicocele that required a varicocelectomy. Using a computerized process, the patients were prospectively randomized into two groups (1:1 ratio, 30 patients each group). Nitroglycerin was administered as a vasodilator during subinguinal loupe-assisted varicocelectomy (LV) in Group A. Subinguinal microscopic varicocelectomy (MV) was performed on Group B. All patients gave their informed consent in compliance with the guidelines set forth by the Fayoum University Faculty of Medicine's ethical committee.

G*Power version 3.1.7 was used to calculate the sample size. In order to reach a power level of 0.80 at an alpha level of 0.05 (two-tailed), a minimum of 20 patients per group were first determined. A power level of 0.95 was attained by increasing the sample size to 30 patients per group to account for possible loss to follow-up. Patients with clinically evident varicocele who presented with primary or secondary infertility, intractable pain, aberrant semen values, and diminished testicular volume were included in the study. The patients ranged in age from 18 to 50. Those with systemic conditions that impact arterial flow, such as diabetes, hypertension, liver disease, and hypercholesterolemia, were excluded if they were younger than 18 or older than 50.

Additionally, patients with subclinical varicocele who had previously had varicocelectomy or inguinoscrotal surgery on the same side were not included.

Every patient had a comprehensive evaluation that included a complete general, local, and genital examination as well as a detailed medical and surgical history.Prior to intervention, all patients underwent two semen analyses. Patients with severe oligospermia and azoospermia underwent hormonal analysis, and routine laboratory tests were performed prior to surgery.

Scrotal ultrasonography and color doppler ultrasonography were used in the radiological examination to measure the resistive index (RI) for the intra-testicular and capsular arteries, show the diameter of the sprematic vein, and assess the degree of reflux using the valsalva maneuver. Doppler and ultrasound evaluations were performed prior to and three months following the surgery

Operative Technique Every patient had a subinguinal varicocelectomy while under general or spinal anesthesia, when needed. Group B used a surgical microscope with ×10 to ×12 magnification, while Group A used a surgical loop (Sinirgia 3.3X expandable field) with the instillation of 1 ml nitroglycerine following the identification and incision of spermatic fascia of the cord for accurate identification of spermatic arteries and veins and prior to vein ligation. recording the entire duration of the procedure, from skin incision to closure. It was noted how many veins were ligated both inside and outside the cord. Vital sign monitoring was done during the process. Evaluation for bleeding, scrotal hematoma, and length of hospital stay were all part of postoperative surveillance. Following surgery, patients were monitored for three months. Repeat semen analysis and a scrotal Doppler evaluation three months after the intervention were part of the follow-up.

Analysis of Statistics

Statistical Analysis After the data was coded and imported into Microsoft Excel, SPSS version 29 for Windows was used for analysis. Counts, percentages, means with standard deviations for parametric data, and medians with ranges for non-parametric data were examples of descriptive statistics. The one-sample Kolmogorov-Smirnov test was used to determine whether quantitative data was normal. The Chi-square test was used to compare nominal qualitative groups, the Mann-Whitney U test was used to compare ordinal qualitative groups, the independent samples t-test was used to compare quantitative measures between independent groups, the paired t-test was used to compare dependent quantitative data, and statistical significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically evident varicocele who presented with primary or secondary infertility
* intractable pain
* aberrant semen values
* and diminished testicular volume were included in the study.

Exclusion Criteria:

* Those with systemic conditions that impact arterial flow, such as diabetes, hypertension, liver disease, and hypercholesterolemia
* Younger than 18 or older than 50.
* Patients with subclinical varicocele
* patients had previously had a varicocelectomy or inguinoscrotal surgery on the same side were not included.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
percent of sperm motility in semen analysis | 3 months
  percent of improvement of sperm motility

SECONDARY OUTCOMES:
testicular Doppler parameters, mainly percentages of resistive index changes | From enrollment to the end of treatment at 12 weeks
  percentages of changes in resistive index in testes

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud Dogha, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
participant request